CLINICAL TRIAL: NCT00214032
Title: Treatment of Arm Lymphedema in Breast Cancer Survivors: A Double-Blind, Randomized Study of Pycnogenol vs. Placebo
Brief Title: Pycnogenol for the Treatment of Lymphedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-0047; NCCAM R21 A1724-01; CC 05302
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-01

CONDITIONS: Lymphedema
Keywords: lymphedema of the arm in breast cancer survivors
MeSH Terms: conditions — Lymphedema | interventions — pycnogenols

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): pycnogenol daily
  Interventions: Drug: Pycnogenol
- 2 (Placebo Comparator): placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pycnogenol — pycnogenol 300 mg daily
  Arms: 1
Drug: Placebo — placebo 3 capsules daily
  Arms: 2

SUMMARY:
The objectives of this study are to evaluate the effectiveness of Pycnogenol (French maritime pine bark extract) for arm lymphedema in women following treatment for breast cancer, to evaluate the accuracy and sensitivity of bioelectric impedence as a measurement of lymphedema of the arm, and to validate the proposed arm lymphedema quality-of-life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months from last surgical and/or radiation treatment to the affected axilla
* Unilateral lymphedema of the upper extremity

Exclusion Criteria:

* May not be receiving or be scheduled to receive cytotoxic or radiation chemotherapy treatment while on this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-05; Primary Completion 2006-11 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
reduction of arm lymphedema | monthly

SECONDARY OUTCOMES:
comparison/validation of bioelectric impedance to measure lymphedema changes, validation of lymphedema questionnaire | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Hutson, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States